CLINICAL TRIAL: NCT05800795
Title: Evaluation of Soft Tissue Response to Titanium Healing Abutments Treated by Erbium: YAG Laser or Plasma Spray: A Randomized Controlled Clinical Study With Histological, and Scanning Electron Microscopic Analysis
Brief Title: Evaluation of Soft Tissue Response to Titanium Healing Abutments Treated by Erbium: YAG Laser or Plasma Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dalia Yosri, Assistant lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecID021817
Record Dates: First submitted 2023-03-05; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Peri-implant Mucositis
Keywords: healing abutment; plasma spray; Er: YAG laser
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: comparison between three groups
Who Masked: Outcomes Assessor
Masking Description: assessor of clinical parameters, histological samples and scanning electron microscopy samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- laser group (Active Comparator): Healing abutments have been treated by Er:YAG laser. The laser-machine (with a wavelength of 2.940 nm) was used with settings of 100 mJ/pulse (12.7 J/cm₂) and 10 Hz. The healing abutments' surface was thoroughly decontaminated by the fiber tip in a semicircular contact mode with copious water irrigation.
  Interventions: Device: Er: YAG laser
- plasma group (Active Comparator): Healing abutments have been sprayed with an atmospheric pressure plasma device (Piezobrush® PZ2)
  , by using active gas, low-temperature plasma treatment under irradiation at 0.2 MPa for a total of 80 seconds at 10 mm (20 seconds per each surface)
  Interventions: Device: plasma spray
- control group (No Intervention): Healing abutments were installed as they came from industry and received no further treatment.

INTERVENTIONS:
Device: Er: YAG laser — surface treatment with Er: YAG laser for heating abutments
  Arms: laser group
Device: plasma spray — surface treatment with plasma spray for heating abutments
  Arms: plasma group

SUMMARY:
The attachment of peri implant soft tissue to the implant serves as a biological seal that can prevent the development of inflammatory peri-implant diseases. Presence of contaminants has been suggested to be associated with tissue damaging inflammation and titanium wear microparticles were demonstrated to activate osteoclastic action. Er: YAG laser has been extensively investigated clinically for applications for treating periimplantitis either independently or in combination with other techniques, showing favorable outcomes. Plasma spray treatment can decontaminate surfaces without modifying their topography. It is also able to increase the surface energy by obtaining more hydrophilic surfaces, which may increase the capacity of the titanium oxide layer to interact with cells and proteins of surrounding tissue improving cell adhesion to the treated surface.

DETAILED DESCRIPTION:
This study was conducted on 24 patients seeking implant placement. A total number of 33 healing abutments were included in this study, they were divided into 3 groups. Group 1 (Laser group): 8 patients in this group received 11 healing abutments treated with Er:YAG laser, group 2 (Plasma group): 8 patients in this group received 11 healing abutments treated with plasma sprayand group 3 (control group): 8 patients in this group received 11 healing abutments with no surface treatment.Three months after implants placement, patients included in the study were randomly assigned to one of the three study groups, second stage surgery was performed and patients received healing abutments without surface treatment in control group, surface treatment was performed in plasma and laser groups. After two weeks, clinical assessment was done using PI and GI before taking biopsies from peri-implant soft tissue for histological assessment. H&E stain was used for measuring inflammatory cells count and Masson's Trichrome stains for measuring collagen fibers area fraction. Analysis of the abutments surface was done using SEM.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age range from 20 to 45 years old.
* Patients need placement of fixed implant-supported prosthesis in maxillary arch.
* Patients who are medically free from any systemic diseases as evidenced by the health questionnaire, using modified Cornell medical index (Pendleton et al., 2004).
* patients with good oral hygiene (Plaque Index and bleeding on probing less than or equal to grade 1).
* Absence of any local conditions affecting bone-implant osseointegration (e.g., infection and poor bone density).
* The presence of sufficient bone width and height that permit the placement of implant with minimum diameter 3.5 mm and 8.5 mm length.

Exclusion Criteria:

* Presence of acute infections.
* Smokers.
* Pregnancy and lactation.
* Patients with a history of bisphosphonates therapy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
histological assessment measuring inflammatory cells count. | two weeks after stage two surgery
  sections of biopsies from peri-implant soft tissue stained with hematoxylin and eosin stain.
  H&E stain was used for measuring inflammatory cells count and Masson's Trichrome stains for measuring collagen fibers area fraction.
histological assessment measuring collagen fibers area fraction. | two weeks after stage two surgery
  sections of biopsies from peri-implant soft tissue stained with Masson trichrome stain.

SECONDARY OUTCOMES:
scanning electron microscopic analysis | two weeks after stage two surgery
  Analysis of the abutments surface was done using SEM
clinical assessment measuring plaque index | two weeks after stage two surgery and after three months
  Clinical assessment was done using loe and silness plaque index score from 0 to 3
clinical assessment measuring gingival index | two weeks after stage two surgery and after three months
  Clinical assessment was done using loe and silness gingival index score from 0 to 3

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University -Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No